CLINICAL TRIAL: NCT05987683
Title: The Efficacy of Thread Embedding Acupuncture on Pain Score, Neck Disability Index, and Pressure Pain Threshold for Myofascial Pain Therapy in the Upper Trapezius Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Emilia Puspitasari Winarno, Doctor, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23060907
Record Dates: First submitted 2023-07-26; First posted 2023-08-14 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Myofascial Pain of Upper Trapezius Muscle

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thread-Embedding Acupuncture (Experimental): Thread-Embedding Acupuncture using a 29-gauge TEA needle with a 50-mm PDO (polydioxanone) thread
  Interventions: Procedure: Thread-Embedding Acupuncture, Sham Thread-Embedding Acupuncture
- Sham Thread-Embedding Acupuncture (Sham Comparator): Sham Thread-Embedding Acupuncture using a 29-gauge TEA needle but thread-removed, just needle alone
  Interventions: Procedure: Thread-Embedding Acupuncture, Sham Thread-Embedding Acupuncture

INTERVENTIONS:
Procedure: Thread-Embedding Acupuncture, Sham Thread-Embedding Acupuncture — Thread-Embedding Acupuncture: using a 29-gauge TEA needle with a 50-mm PDO (polydioxanone) thread Sham Thread-Embedding Acupuncture: using a 29-gauge TEA needle but thread-removed, just needle alone

SUMMARY:
Myofascial pain is characterized by myofascial trigger points, considered as a major cause of neck and shoulder pain in the working population. Thread-embedding acupuncture is a new acupuncture modality that can provide long-term stimulation aimed at prolonging its therapeutic effect that is similar to conventional acupuncture, such as analgesic effects. The goal of this randomized controlled trial is to evaluate and compare the effects of thread-embedding acupuncture and sham thread-embedding acupuncture as a therapy for myofascial pain in the upper trapezius muscle. The primary aim of this study is to investigate whether thread-embedding acupuncture therapy gives better and last longer results for myofascial pain of the upper trapezius muscle than sham thread-embedding acupuncture.

DETAILED DESCRIPTION:
This is a clinical trial study to evaluate and compare the effects of thread-embedding acupuncture and sham thread-embedding acupuncture as a therapy for myofascial pain in the upper trapezius muscle. The subjects are 44 males/female with myofascial pain in the upper trapezius muscle and will be randomly assigned to 2 groups: (1) thread-embedding acupuncture and (2) Sham thread-embedding acupuncture. The subjects will receive a single treatment. The outcome will be assessed before treatment (baseline) and 3 days, 1 week, 4 weeks, 8 weeks after treatment. Patients and the outcome assessors will be blinded to the group allocation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-59 years.
* Subject with myofascial pain in the upper trapezius muscle.
* VAS score of 30-70 mm from 100 mm during activities (everyday activities or light exercise).
* Pain > 3 months.
* Willing to participate in this research to completion and sign informed consent.

Exclusion Criteria:

* Fibromyalgia.
* Have had cervical spine surgery.
* Have done Dry needling therapy on the upper trapezius muscle in the last 9 days
* Have done thread acupuncture on the upper trapezius muscle in the last 6 months.
* Have performed pharmacopuncture on the upper trapezius muscle in the last 6 months.
* VAS score is more than 70 mm than 100 mm at resting.
* History of anti-inflammatory drug treatment in the previous 2 weeks.
* History of intra-articular steroid injections in the previous 3 months.
* There is a tumor, wound, or skin infection at the needle insertion area.
* Fever (≥ 37.5 oC).
* There is a hypersensitivity reaction in previous acupuncture therapy (metal allergy, severe atopy, keloids, or other skin hypersensitivity).
* Suffering from a blood disorder or taking blood thinners (anti-platelet or anti-coagulant drugs).
* Have a heart condition or uncontrolled diabetes.
* Blood glucose level (GDS) ≥200 mg/dL is checked by capillary blood using a glucometer.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2023-08-21 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | before treatment (baseline) and 3 days, 1 week, 4 weeks, 8 weeks after treatment
  Pain rating scale for measuring pain

SECONDARY OUTCOMES:
Neck Disability Index | before treatment (baseline) and 3 days, 1 week, 4 weeks, 8 weeks after treatment
  A questionnaire for measuring self-rated disability due to neck pain
Pressure Pain Threshold | before treatment (baseline) and 3 days, 1 week, 4 weeks, 8 weeks after treatment
  Using the minimum force applied which induces pain, measured with algometer

CONTACTS AND LOCATIONS:
Overall Officials: KEPK FKUI-RSCM, Principal Investigator — The Ethics Committee of the Faculty of Medicine, University of Indonesia - Cipto Mangunkusumo Hospital
Locations (2):
- Indonesia (2):
  - Cipto Mangunkusumo Hospital, Jakarta, DKI Jakarta
  - Persahabatan Hospital, Jakarta, DKI Jakarta

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol